CLINICAL TRIAL: NCT01302652
Title: Effects of Physiologic Growth Hormone Administration on Echocardiographic Parameters in Subjects With Growth Hormone Deficiency Following Cure of Acromegaly
Brief Title: Effect of Growth Hormone (GH) on Cardiac Echos in GH Deficient Patients After Acromegaly Treatment
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2010P002188
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Acromegaly
Keywords: acromegaly; growth hormone; growth hormone deficiency
MeSH Terms: conditions — Acromegaly; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GH deficient after acromegaly cure (on GH replacement): Men and women with growth hormone deficiency following cure of acromegaly who are receiving growth hormone treatment.
- GH deficient after acromegaly cure (not on GH replacement): Men and women with growth hormone deficiency following cure of acromegaly who are not receiving growth hormone treatment.

SUMMARY:
The purpose of this research study is to study the effects of growth hormone (GH) replacement on the heart. The investigators will study these effects in people who have been cured of acromegaly and then have developed growth hormone deficiency (GHD, not enough growth hormone).

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* history of acromegaly with biochemical cure
* growth hormone deficiency

Exclusion Criteria:

* untreated thyroid disease within the past 3 months
* untreated adrenal insufficiency within the past 3 months
* uncontrolled hypertension
* congestive heart failure
* gonadal steroid therapy within the past 3 months
* pregnancy or nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women between age 18-75 who have developed growth hormone deficiency after history of acromegaly with biochemical cure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Echocardiographic Findings at One Year | baseline and one year

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States